CLINICAL TRIAL: NCT07117214
Title: A Phase I, Open Label First in Human Study to Evaluate the Imaging Performance, Safety, Biodistribution and Pharmacokinetics of [68Ga]Ga-DWJ155 in Adult Patients With Advanced Breast Cancer and Advanced NSCLC
Brief Title: A Phase I Study of [68Ga]Ga-DWJ155 in Patients With Breast and Lung Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CFKL480A02101; 2024-517746-34 (Other: EU CTIS number)
Record Dates: First submitted 2025-07-22; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Breast cancer; Non-small cell lung cancer; Radioligand imaging; [68Ga]Ga-DWJ155; FKL480; gallium; adenocarcinoma; ductal; lobular; positron emission tomography (PET); dosimetry
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced breast cancer (Experimental): Patients will receive FKL480 ([68Ga]Ga-DWJ155)
  Interventions: Drug: [68Ga]Ga-DWJ155
- Advanced NSCLC (Experimental): Patients will receive FKL480 ([68Ga]Ga-DWJ155)
  Interventions: Drug: [68Ga]Ga-DWJ155

INTERVENTIONS:
Drug: [68Ga]Ga-DWJ155 — Radioligand imaging agent

SUMMARY:
This is a phase I, open label first in human study to evaluate the imaging performance, safety, biodistribution and pharmacokinetics of [68Ga]Ga-DWJ155 in patients ≥ 18 years of age with hormone receptor positive/HER2 negative (HR+/HER2-) and HER2 positive (HER2+) advanced breast cancer (aBC) and advanced Non-Small Cell Lung Cancer (aNSCLC) adenocarcinoma.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), open-label, phase I radioligand imaging study designed to assess the biodistribution, imaging, safety, PK and dosimetry properties in patients with aBC and aNSCLC adenocarcinoma.

Approximately 15-21 aBC and 9-15 aNSCLC patients will be enrolled into the study. All patients enrolled in the study will receive a single administered radioactive dose of FKL480. The study will consist of an imaging characterization part and an expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with histologically or cytologically confirmed and documented HR+/HER2- advanced breast cancer (aBC), advanced defined as locoregionally advanced unresectable or metastatic, either untreated or currently receiving first line of systemic therapy OR patients with histologically or cytologically confirmed and documented HER2+ aBC, advanced defined as locoregionally advanced unresectable or metastatic, either untreated or relapsed/refractory (r/r) after one or more lines of treatment OR patients with histologically or cytologically confirmed and documented advanced NSCLC (aNSCLC) adenocarcinoma, advanced defined as locoregionally unresectable or metastatic, either untreated or currently receiving first line of systemic therapy.
* Presence of measurable disease (at least one target lesion) according to RECIST v1.1 assessed by conventional CT scan.

Exclusion Criteria:

* Patients having out of range laboratory values for kidney function and blood markers as defined in the study protocol
* Patients with inadequate hepatic function
* Unmanageable urinary tract obstruction or urinary incontinence

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Standard Uptake Value (SUV) mean and max of FKL480 uptake in normal organs and tumor lesions over time | Up to 240 minutes after dosing on Day 1
  Imaging properties of FKL480 will be evaluated by assessing radiotracer uptake, identified via positron emission tomography (PET) scans. The SUVmean and SUVmax will be calculated and reported with summary statistics.
Standard Uptake Value ratio (SUVr) of FKL480 uptake in normal organs and tumor lesions over time | Up to 240 minutes after dosing on Day 1
  SUVr will be calculated by dividing the SUV of the lesions by the SUV of the different organs in order to identify the reference organ with the lowest uptake and the respective SUVr (i.e. using SUVmean or SUVmax).

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 3 days after single dose administration on Day 1
  Incidence and severity of AEs and SAEs, including changes in vital signs and laboratory values qualifying and reported as AEs.
Dosimetry sub-group: Observed maximum concentration (Cmax) of FKL480 based on blood radioactivity data | Up to 240 minutes after dosing on Day 1
  The FKL480 pharmacokinetic analysis will be performed based on blood radioactivity concentration data, obtained by measuring in gamma-counting equipment the blood samples.
Dosimetry sub-group: Observed area under the curve (AUC) from time zero to the last measurable concentration sampling time (AUClast) of FKL480 based on blood radioactivity data | Up to 240 minutes after dosing on Day 1
  The FKL480 pharmacokinetic analysis will be performed based on blood radioactivity concentration data, obtained by measuring in gamma-counting equipment the blood samples
Dosimetry sub-group: Observed time to reach maximum (Tmax) after single dose administration of FKL480 based on blood radioactivity data | Up to 240 minutes after dosing on Day 1
  The FKL480 pharmacokinetic analysis will be performed based on blood radioactivity concentration data, obtained by measuring in gamma-counting equipment the blood samples
Dosimetry sub-group: Urinary excretion of FKL480 | Up to 240 minutes after dosing on Day 1
  The elimination of the compound in urine will be evaluated based on urine radioactivity concentration data obtained by measuring in gamma counting equipment the urine samples.
Dosimetry sub-group: Absorbed radiation dose in normal tissues and total body | Up to 240 minutes after dosing on Day 1
  Absorbed radiation dose coefficients in selected organs and lesions and total body as measured by image quantification.
Dosimetry sub-group: Effective dose | Up to 240 minutes after dosing on Day 1
  Effective dose in selected organs and total body as measured by image quantification.

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.